CLINICAL TRIAL: NCT02795975
Title: Clinical Evaluation of the Aptima® Combo 2® Assay Using the Panther® System in Female Urine Samples
Status: Terminated | Type: Observational
Why Stopped: Sponsor business decision
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A10417-AC2PS-CSP-02
Record Dates: First submitted 2016-06-02; First posted 2016-06-10 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Chlamydia Trachomatis; Gonorrhea
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the performance characteristics of the AC2 assay on the Panther system using female urine specimens.

ELIGIBILITY:
Inclusion Criteria:

* The subject is ≥14 years of age at the time of enrollment and is currently sexually active (eg, has had penile/vaginal intercourse within the past 6 months).
* For subjects under 18 years old, assent of the subject and/or parental/legal guardian permission has been obtained if required by the institutional review board (IRB).
* The subject and/or legally authorized representative is willing and able to undergo the informed consent process prior to study participation, and:
* reports symptoms consistent with a suspected STI (eg, abnormal discharge, genital itching, pain/discomfort during sexual intercourse or urination, and/or lower abdominal discomfort); or
* is asymptomatic and known to be partners with, or a contact of, a person with a confirmed or suspected STI; or
* is asymptomatic and undergoing screening evaluation for possible STIs; or
* is asymptomatic and undergoing a routine pelvic examination.

Exclusion Criteria:

* The subject took antibiotic medications within the last 21 days prior to collection.
* The subject already participated in the study.
* The subject has a history of illness that the PI or designee considers could interfere with or affect the conduct, results, and/or completion of the study.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sexually active women ≥14 years of age with or without symptoms of STIs will be eligible for enrollment. Participating clinical collection sites may include US family planning, public health, and STI clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1766 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | Enrollment ongoing until estimated March 2017

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Planned Parenthood of Southern New England, Inc, New Haven, Connecticut
  - Segal Institute for Clinical Research, Miami, Florida
  - Eskenazi Hospital - Indiana University School of Medicine, Indianapolis, Indiana
  - Clinical Trials Management, LLC, Mandeville, Louisiana
  - Beyer Research, Kalamazoo, Michigan
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - LabCorp, Burlington, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Multnomah County Health Department, STD Clinic, Portland, Oregon
  - Geneuity, Maryville, Tennessee
  - Planned Parenthood Gulf Coast, Inc., Houston, Texas
  - Brownstone Clinical Trials, Irving, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Tidewater Clinical Research, Inc., Virginia Beach, Virginia
  - University of Washington Center for AIDS & STD, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No